CLINICAL TRIAL: NCT05055804
Title: The ELG Analysis of Glucose a Correlational to Blood Glucose Assa
Brief Title: The ELG Analysis of Glucose a Correlational to Blood Glucose Assay
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: XP Technology, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Q151642/S001
Record Dates: First submitted 2021-09-01; First posted 2021-09-24 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: ELG; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ELG Device Comparison to Whole Blood Testing (Experimental): Participant will place thumb in the ELG device for scan. Scan generally takes between 1-2 minutes. ELG then displays a readout of both a glucose and A1C reading on the screen of the ELG device.
  Interventions: Device: ELG

INTERVENTIONS:
Device: ELG — The effectiveness of ELG to standardized blood test methods (fingerstick) and comparison to AlcNOW + (or equivalence) and of laboratory test results.
  Human subject requirements during ELG study will not challenge diabetics or non-diabetics glycemic event. For example, diabetes type 1, the subject will not have to adjust their insulin or glucose. For type 2 diabetes, the subject will not have to adjust their oral hypoglycemic agent or glucose, as well.
  Other Names: ELG, Easy Light Glycometer

SUMMARY:
This study is an investigational study of the ELG medical device to monitor glucose blood level in diabetes mellitus Type 1 and 2 without blood samples in comparison to blood testing methods."Investigational" means the ELG medical device is subjected by the FDA (Food and Drug Administration) for premarket testing requirements. The purpose of this study is to collect data comparison values between ELG testing device to current blood testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 1 or 2 diabetes
* Be 25 - 65 years of age
* Male or female
* Various ethnicities are desired
* Must be available for 2 visits within a 2-4 week period and willing to spend up to 1-2 hours/visit
* Must have daytime availability for visits
* Able to have 1 venous blood draw & up to 4 fingersticks for complete blood testing at each visit
* Must be willing and able to fast (for at least 6 hours) prior to first visit

Exclusion Criteria:

* Taking drugs of abuse (illegal and/or prescription)
* Have been in another research study in the last 30 days
* Have had a blood transfusion or severe blood loss in the last 14 days
* Have Sickle Cell Anemia

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Standard OTC Glucose, A1C & Laboratory Results in Comparison to ELG Device During Fasting Event | Visit will last for up to 1-2 hours. This outcome will measure overnight fasting results.
  Measuring precision and accuracy of ELG (glucose/A1C %) without blood samples, by performance evaluation to 3 different standard OTC fingerstick, A1C Now (or equivalent OTC brand) and NGSP-certified lab, using whole blood comparative tests with use of venous blood draw/fingersticks and NGSP-certified lab, and assess confidence limits to Bland-Altman plot, after overnight fasting for a minimum of 6 hours.
Standard OTC Glucose, A1C & Laboratory Results in Comparison to ELG Device During Non-Fasting Event | This visit will be measured within a 4 week time frame, following the 1st visit. This visit will last for up to 1-2 hours. This outcome will measure non-fasting results.
  Measuring precision and accuracy of ELG (glucose/A1C %) without blood samples, by performance evaluation to 3 different standard OTC fingerstick, A1C Now (or equivalent OTC brand) and NGSP-certified lab, using whole blood comparative tests with use of venous blood draw/fingersticks and NGSP-certified lab, and assess confidence limits to Bland-Altman plot, during non-fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joe P Rouse, MD, Principal Investigator; Dr. Peter P Xaysanasy, DPM, Study Director — XP Technology, LLC
Locations (1):
- Rouse Family Medical Clinic, Springdale, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No